CLINICAL TRIAL: NCT02672241
Title: Phase 2 Study of Nimotuzumab in Combination With Radio-chemotherapy for the Treatment of Brainstem Tumor in Children
Brief Title: Nimotuzumab in Combination With Radio-chemotherapy for the Treatment of Brainstem Tumor in Children
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Chuanying Zhu, doctor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sanghaixinhua-002
Record Dates: First submitted 2016-01-31; First posted 2016-02-03 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Childhood Brain Stem Neoplasm
Keywords: Radiation Therapy; Brainstem Tumor in Children
MeSH Terms: interventions — nimotuzumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- radio-chemotherapy plus nimotuzumab (Experimental): Radiotherapy: The total radiation dose is 52.2Gy (1.8Gy fractions). Chemotherapy: Nimotuzumab, given during radiotherapy, is administered via intravenous drip with a dosage of 150mg/m2, weekly, for 6 consecutive weeks. After radiotherapy and evaluation, disease progression-free patients will continue to receive Nimotuzumab treatment biweekly until disease relapse or progression. Temozolomide is applied to these patients as a chemotherapy drug with a dosage of 75mg/m2, daily. The chemotherapy and radiation therapy are combined as temozolomide is taken 1 hour prior to every fraction of radiotherapy. In 4 weeks after the completion of radiotherapy, temozolomide is given for 8 cycles.
  Interventions: Drug: Nimotuzumab; Drug: Temozolomide

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab given during radiotherapy, is administered via intravenous drip with a dosage of 150mg/m2, weekly, for 6 consecutive weeks. After radiotherapy and evaluation, disease progression-free patients will continue to receive Nimotuzumab treatment biweekly until disease relapse or progression.
  Other Names: h-R3, BIOMAb EGFR, Biocon
Drug: Temozolomide — Temozolomide is applied to these patients as a chemotherapy drug with a dosage of 75mg/m2, daily. The chemotherapy and radiation are combined as temozolomide is taken 1 hour prior to every fraction of radiotherapy. In 4 weeks after the completion of radiotherapy, temozolomide is given for 8 cycles (dosage: the 1st cycle, 150mg/m2, daily × 5 days, 4 weeks a cycle; the 2-8th cycle, 200mg/m2, daily × 5 days, 4 weeks a cycle and repeated again).
  Other Names: brand names Temodar and Temodal and Temcad

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of nimotuzumab in combination of radio-chemotherapy for the treatment of brainstem tumor in children.

DETAILED DESCRIPTION:
Nimotuzumab (h-R3), a recombinant humanized monoclonal immunoglobulin G1 antibody that binds to the extracellular domain of EGFR, which blocks the binding of EGF and transforming growth factor-α to EGFR. High expression of EGFR protein in glioma has been associated with tumor progression and enhanced tumorigenicity. Several clinical trials have demonstrated the anti-tumor effects of nimotuzumab, such as head and neck cancer and esophageal cancer15. The purpose of this study was to evaluate the efficacy of nimotuzumab in combination of radio-chemotherapy for the treatment of brainstem tumors in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >/= 3 and </= 21 years of age.
* Patients must have a newly diagnosed or progressive brain stem tumor.
* If biopsy has been performed, patients with both high and low grade astrocytomas are eligible.
* Non-histologically confirmed brain stem tumors are eligible. Neuroradiographic confirmation of brain stem glioma is mandatory for study entry.
* Cervicomedullary junction tumors are ineligible.
* Patients with a diagnosis of NF-1 are ineligible.
* Patients must be registered within 6 weeks from diagnosis or recurrence.
* Patients must have life expectancy > 6 weeks.
* Patients must have adequate hematologic and renal function: ANC >1,000/ul, platelets>100,000/ul and creatinine normal for age: </= 0.7 mg/dl (age 3-10yrs.), </= 1.0 mg/dl (11-12yrs.). and </= 1.2 (13-21yrs.).
* Written informed consent must be obtained according to institutional guidelines.

Exclusion Criteria:

* Cervicomedullary junction tumors are ineligible.
* Patients with a diagnosis of NF-1 are ineligible.
* Pregnant or nursing women are ineligible.
* Patients must not start treatment until informed consent is given and the patient is registered.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | first analysis will occur 1 month after accrual of all patients

SECONDARY OUTCOMES:
Progression free survival(PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Objective response rate (ORR) | first analysis will occur 1 month after accrual of all patients

CONTACTS AND LOCATIONS:
Overall Officials: mawei jiang, MD, Principal Investigator — The Department of Radiation Oncology, Xin Hua Hospital affiliated to Shanghai Jiaotong University School of Medicine
Locations (1):
- he Department of Radiation Oncology, Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes